CLINICAL TRIAL: NCT03411655
Title: A Randomised Non Crossover Study Comparing Ambu® Aura-ITM and Ambu® Aura GainTM for Fiberoptic Intubation in Children
Brief Title: Ambu® Aura-ITM Versus Ambu Aura GainTM for Fiberoptic Intubation in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Schulthess Klinik (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Christian Keller, MD M.Sc., Schulthess Klinik
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Schulthess_Anä_13
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambu® Aura-ITM (Active Comparator)
  Interventions: Device: Ambu® Aura-ITM
- Ambu Aura GainTM (Active Comparator)
  Interventions: Device: Ambu Aura GainTM

INTERVENTIONS:
Device: Ambu Aura GainTM — Time and success rate
  Arms: Ambu Aura GainTM
Device: Ambu® Aura-ITM — Time and success rate
  Arms: Ambu® Aura-ITM

SUMMARY:
The investigators test the hypothesis that fiberoptic intubation (time and success rate) differ between the Ambu® Aura-ITM and Ambu Aura GainTM in paralyzed anaesthetized pediatric patients

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* age 1.5 - 6 years
* minor surgery
* extraglottic airway device

Exclusion Criteria:

* age (<18 months, >6 years)
* weight (<10 kg, >20 kg)
* a known difficult airway
* risk of aspiration

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Fiberoptic intubation | 5 minutes
  The airway tube view was scored using an established scoring system (4=only vocal cords visible; 3=vocal cords plus posterior epiglottis; 2=vocal cords plus anterior epiglottis; 1=vocal cords not seen)

IPD SHARING:
Plan to Share IPD: No